CLINICAL TRIAL: NCT06567379
Title: Evaluation of Right Ventricular Myocardial Work in Patients With Pulmonary Arterial Hypertension
Brief Title: Myocardial Work Evaluation in Patients With PAH
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2024PI
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAH patients: Patients with heritable, idiopathic PAH or PAH associated with portal hypertension or with drugs.

SUMMARY:
Right ventricular function is a key determinant of survival in patients with pulmonary arterial hypertension, with right heart failure being the leading cause of death. ERS/ESC guidelines recommend evaluating RV function at diagnosis and at first reevaluation under treatment to estimate the one-year mortality risk. However, few RV function markers address both systolic function and afterload. Noninvasive myocardial work is a promising new tool that incorporates systolic function and its afterload into global longitudinal strain. Initially developed for the left ventricle, it can be adapted for the RV using pressure-strain loops. The article aims to evaluate the association of RV myocardial work parameters with the estimate one-year mortality in patients with PAH.

This retrospective study will include patients diagnosed with PAH with transthoracic echocardiography and right heart catheterization within 48 hours at diagnosis and first reevaluation. Patients with unanalyzable echocardiography data will be excluded.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare hemodynamic disease characterized by pre-capillary pulmonary hypertension (PH), due to pulmonary vascular remodeling. Despite the recent development of effective therapies, right ventricular (RV) function remains a key determinant of survival as right heart failure remains the main cause of death among patients with PAH. According to ESC/ERS guidelines, RV function should be evaluated in patients with PAH at baseline (by echocardiography or cardiac MRI) to assess one-year mortality risk, thereby impacting on patient treatment. However, few RV function markers address both the systolic function of the RV and its afterload (i.e., RV-pulmonary artery coupling), which seems necessary in PAH, where the disease is characterized by a progressive increase in pulmonary artery pressures and subsequently, an alteration in RV systolic function. Noninvasive myocardial work is a promising new tool for the evaluation of RV systolic function developed to help differentiate reduced myocardial performance due to increased afterload versus reduced myocardial contractibility. It was first developed for left ventricular assessment but can be adapted to the RV using pressure-strain loops. Very few data on its use on RV function are available but the results are promising. However, its value in patients with PAH and its evolution after PAH treatment initiation has never been evaluated. Thus, the aim of this article is to evaluate the association of RV myocardial work parameters at baseline and at first reevaluation with estimated one-year mortality risk in patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive incident patients with a diagnosis of idiopathic, heritable, drug-associated PH, or associated with portal hypertension and referred to PH reference center in Nancy university hospital.
* Transthoracic echocardiography (TTE) and a right heart catheterization (RHC) within 48 hours at diagnosis and at first reevaluation with PAH treatment

Exclusion Criteria:

* cardiac ultrasound data not analyzable (poor echogenicity or poor quality of RV slice). - -- Patients with PH associated with left-heart disease (group 2), PH associated with lung diseases and/or hypoxia (group 3), PH associated with pulmonary artery obstructions (group 4) and PH with unclear and/or multifactorial mechanisms (group 5) were also excluded. Patients with a positive response to the vasoreactivity test or with features of venous or capillaries involvement were also excluded.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PAH patients referred to PH reference center in Nancy university Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
One year risk mortality | six months
  According to four model strata, estimation of one year mortality risk (low, intermediate-low, intermediate-high or high risk)

CONTACTS AND LOCATIONS:
Locations (1):
- Valentin, Nancy, France

IPD SHARING:
Plan to Share IPD: No